CLINICAL TRIAL: NCT00751777
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Immunogenicity and Safety of a Two Vaccination Regimen With an LT Vaccine Patch in Healthy Adults
Brief Title: Traveler's Diarrhea (TD) Automated Process
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ELT207
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Prevention of Travelers' Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: 37.5 µg LT patch (Experimental): 80 subjects will receive a two vaccination regimen with a LT patch.
  Interventions: Biological: heat-labile enterotoxin of E. coli (LT)
- Group 2: 0 µg LT patch (placebo) (Placebo Comparator): 40 subjects will receive a two vaccination regimen with a placebo patch.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: heat-labile enterotoxin of E. coli (LT) — Travelers' Diarrhea Vaccine System
  Other Names: TD Vaccine System
  Arms: Group 1: 37.5 µg LT patch
Biological: Placebo — Travelers' Diarrhea Vaccine System
  Other Names: TD Vaccine System
  Arms: Group 2: 0 µg LT patch (placebo)

SUMMARY:
To evaluate and compare the immune responses and safety following a two vaccination regimen by transcutaneous immunization with heat-labile enterotoxin of E. coli (LT) patches or placebo patches.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females, 18-64 years of age (inclusive) at the planned start of the study (first vaccination on Day 0)
* Signed Informed Consent
* Women who are not post-menopausal or surgically sterile must have a negative serum/urine pregnancy test at screening and within 24 hours of each vaccination with understanding (through Informed Consent process) to not become pregnant and to employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: abstinence, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom or diaphragm, with spermicide), and IUD.

Exclusion Criteria:

* Laboratory abnormalities [as determined by the Toxicity Grading Scale (grade 1 4)] at laboratory screening
* Abnormalities at physical examination [as determined by the Toxicity Grading Scale (grade 1-4)]
* Known allergies to any component of the vaccine
* Known allergies to adhesives
* Participated in research involving investigational product within 30 days before planned date of first vaccination or within 90 days after first vaccination
* Donated blood or blood products such as plasma within 30 days prior to planned date of first vaccination or within 90 days after first vaccination
* Ever received investigational enterotoxigenic E. coli, LT, or LT (R192G) or NasalFlu, Berna Biotech, Ltd
* Ever received cholera toxin or vaccine (e.g. Orochol™, Dukoral™)
* History of diarrhea while traveling in a developing country within the last year
* History of abdominal surgery (excluding C-section, hysterectomy, cosmetic surgery, liposuction, appendectomy, cholecystectomy, ventral hernia repair, and other surgeries not pertaining to gastrointestinal problems) or history of, or recent acute gastrointestinal illness
* Positive serology for HIV-1, HIV-2, HBsAg, or HCV
* Medical history of acute or chronic skin disease at vaccination area(s)
* Active skin allergy
* Signs of acute skin infection, sunburn or skin abnormalities at the vaccination area(s) including fungal infections, severe acne, or active contact dermatitis, or a history of keloid formation
* Excessively hirsute and unwilling to clip hair at the vaccination area(s)
* Visible tattoos or marks (tattoos/scars) at the vaccination area(s) that would prevent appropriate dermatologic monitoring of the vaccination site(s)
* Fever greater than or equal to 38.0°C (100.4°F) at the time of planned vaccination
* Women who are pregnant or breastfeeding
* Acute illness at screening and unresolved at time of planned vaccination
* Employee of the investigational site

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Research Associates
Locations (3):
- United States (3):
  - Solano Clinical Research, Vallejo, California
  - Miami Research Associates, South Miami, Florida
  - Clinical Trials of Texas, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: 37.5 µg LT Patch | Group 2: 0 µg LT Patch (Placebo)
Started | 81 | 39
Completed | 70 (Day 380: study completion for LT group) | 36 (Day 194: study completion for placebo group)
Not Completed | 11 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all study subjects who were consented, randomized, and had a baseline serology
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 37.5 µg LT Patch | Group 2: 0 µg LT Patch (Placebo) | Total
Number analyzed (Participants) | 81 | 39 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.2) | 35.3 (13.0) | 34.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 26 | 72
  Male | 35 | 13 | 48

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) After First and Second Vaccination With LT Vaccine Patch and Comparison Against Placebo
Time Frame: Day 0, Day 14, Day 21, Day 28, Day 35, Day 90, Day 194
Population: Immunogenicity Evaluable Population (IEP): all study subjects who are consented, randomized, received the assigned treatments (both vaccinations), and had blood drawn for immunogenicity testing at baseline (Day 0) and both of the following time points: Day 21 and Day 35.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group 1: 37.5 µg LT Patch | Group 2: 0 µg LT Patch (Placebo)
Number analyzed (Participants) | 76 | 34
geometric mean titer
  GMT LT IgG - Day 0 | 432.6 [349.0 to 536.2] | 400.5 [290.5 to 552.2]
  GMT LT IgG - Day 14 | 4477.5 [3249.6 to 6169.4] | 490.6 [303.8 to 792.2]
  GMT LT IgG - Day 21 | 9107.7 [6791.9 to 12213.0] | 462.1 [298.0 to 716.6]
  GMT LT IgG - Day 28 | 13411.9 [10420 to 17263.5] | 372.6 [255.4 to 543.4]
  GMT LT IgG - Day 35 | 15024.3 [11893 to 18979.4] | 383.6 [270.5 to 544.0]
  GMT LT IgG - Day 90 | 6823.7 [5553.1 to 8385.1] | 156.2 [114.5 to 213.1]
  GMT LT IgG - Day 194 | 2489.2 [1965.5 to 3152.4] | 100.2 [70.7 to 142.0]
  GMT LT IgA - Day 0 | 49.4 [37.4 to 65.1] | 58.9 [38.9 to 89.1]
  GMT LT IgA - Day 14 | 395.6 [289.9 to 539.8] | 59.1 [37.2 to 94.1]
  GMT LT IgA - Day 21 | 619.2 [466.2 to 822.4] | 60.9 [39.8 to 93.0]
  GMT LT IgA - Day 28 | 780.0 [603.8 to 1007.7] | 53.9 [36.8 to 79.1]
  GMT LT IgA - Day 35 | 681.2 [526.1 to 882.0] | 52.5 [35.7 to 77.3]
  GMT LT IgA - Day 90 | 348.1 [280.3 to 432.4] | 40.5 [29.2 to 56.1]
  GMT LT IgA - Day 194 | 177.0 [145.3 to 215.5] | 32.6 [24.3 to 43.6]

2. Primary Outcome: Geometric Mean Fold Ratio (GMFR) After First and Second Vaccination With LT Vaccine Patch and Comparison Against Placebo
Description: GMFRs relative to the baseline titer were determined at each post-baseline time point. All GMFRs were based on log10-transformed data.
Time Frame: Day 14, Day 21, Day 28, Day 35, Day 90, Day 194
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: 37.5 µg LT Patch | Group 2: 0 µg LT Patch (Placebo)
Number analyzed (Participants) | 76 | 34
ratio
  GMFR LT IgG - Day 14 | 10.4 [7.4 to 14.5] | 1.2 [0.7 to 2.0]
  GMFR LT IgG - Day 21 | 21.1 [15.2 to 29.2] | 1.2 [0.7 to 1.9]
  GMFR LT IgG - Day 28 | 31.0 [23.5 to 41.0] | 0.9 [0.6 to 1.4]
  GMFR LT IgG - Day 35 | 34.7 [26.6 to 45.4] | 1.0 [0.6 to 1.4]
  GMFR LT IgG - Day 90 | 16.0 [12.4 to 20.8] | 0.4 [0.3 to 0.6]
  GMFR LT IgG - Day 194 | 5.7 [4.3 to 7.5] | 0.2 [0.2 to 0.4]
  GMFR LT IgA - Day 14 | 8.0 [5.8 to 11.0] | 1.0 [0.6 to 1.6]
  GMFR LT IgA - Day 21 | 12.5 [9.3 to 16.8] | 1.0 [0.7 to 1.6]
  GMFR LT IgA - Day 28 | 15.8 [12.1 to 20.7] | 0.9 [0.6 to 1.4]
  GMFR LT IgA - Day 35 | 13.8 [10.6 to 17.9] | 0.9 [0.6 to 1.3]
  GMFR LT IgA - Day 90 | 7.1 [5.5 to 9.2] | 0.6 [0.4 to 1.0]
  GMFR LT IgA - Day 194 | 3.4 [2.6 to 4.6] | 0.5 [0.3 to 0.8]

3. Primary Outcome: Seroconversion (SCR) After First and Second Vaccination With LT Vaccine Patch and Comparison Against Placebo
Description: Definition of SCR:
  * Seroconversion IgG: ≥ 2-fold rise of LT IgG titer relative to baseline
  * Seroconversion IgA: ≥ 4-fold rise of LT IgA titer relative to baseline
Time Frame: Day 14, Day 21, Day 28, Day 35, Day 90, Day 194
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: 37.5 µg LT Patch | Group 2: 0 µg LT Patch (Placebo)
Number analyzed (Participants) | 76 | 34
percentage of participants
  SCR LT IgG - Day 14 | 77.6 [66.6 to 86.4] | 8.8 [1.9 to 23.7]
  SCR LT IgG - Day 21 | 89.5 [80.3 to 95.3] | 8.8 [1.9 to 23.7]
  SCR LT IgG - Day 28 | 97.4 [90.8 to 99.7] | 2.9 [0.1 to 15.3]
  SCR LT IgG - Day 35 | 97.4 [90.8 to 99.7] | 5.9 [0.7 to 19.7]
  SCR LT IgG - Day 90 | 98.7 [92.8 to 100] | 9.1 [1.9 to 24.3]
  SCR LT IgG - Day 194 | 83.3 [72.7 to 91.1] | 0 [0 to 10.6]
  SCR LT IgA - Day 14 | 57.9 [46.0 to 69.1] | 0.0 [0.0 to 10.3]
  SCR LT IgA - Day 21 | 71.1 [59.5 to 80.9] | 0.0 [0.0 to 10.3]
  SCR LT IgA - Day 28 | 82.9 [72.5 to 90.6] | 0.0 [0.0 to 10.3]
  SCR LT IgA - Day 35 | 81.6 [71.0 to 89.5] | 2.9 [0.1 to 15.3]
  SCR LT IgA - Day 90 | 68.0 [56.2 to 78.3] | 3.0 [0.1 to 15.8]
  SCR LT IgA - Day 194 | 50.0 [38.0 to 62.0] | 0.0 [0.0 to 10.6]

4. Secondary Outcome: Evaluation of Safety of LT Vaccine Patch After First and Second Vaccination Compared to Placebo Patch
Description: LT subjects (Group 1) were followed for six months longer (until Day 380) than Placebo subjects (Group 2) (until Day 194)
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 37.5 µg LT Patch | Group 2: 0 µg LT Patch (Placebo)
Number analyzed (Participants) | 81 | 39
Participants
  AEs : All AEs - vaccination 1 | 75 | 26
  AEs : All AEs - vaccination 2 | 76 | 24
  AEs : Local AEs - vaccination 1 | 73 | 19
  AEs : Systemic AEs - vaccination 1 | 43 | 18
  AEs : Local AEs - vaccination 2 | 73 | 13
  AEs : Systemic AEs - vaccination 2 | 44 | 18
  Severe AEs : All AEs - vaccination 1 | 2 | 2
  Severe AEs : All AEs - vaccination 2 | 2 | 0
  Severe AEs : Local AEs - vaccination 1 | 0 | 0
  Severe AEs : Systemic AEs - vaccination 1 | 2 | 2
  Severe AEs : Local AEs - vaccination 2 | 0 | 0
  Severe AEs : Systemic AEs - vaccination 2 | 2 | 0
  AEs requiring Treatment : All AEs - vaccination 1 | 24 | 6
  AEs requiring Treatment : All AEs - vaccination 2 | 33 | 10
  AEs requiring Treatment : Local AEs - vacc. 1 | 10 | 0
  AEs requiring Treatment : Systemic AEs - vacc. 1 | 16 | 6
  AEs requiring Treatment : Local AEs - vacc. 2 | 4 | 0
  AEs requiring Treatment : Systemic AEs - vacc. 2 | 31 | 10
  related AEs : All AEs - vaccination 1 | 74 | 20
  related AEs : All AEs - vaccination 2 | 74 | 13
  related AEs : Local AEs - vaccination 1 | 73 | 19
  related AEs : Systemic AEs - vaccination 1 | 17 | 5
  related AEs : Local AEs - vaccination 2 | 73 | 13
  related AEs : Systemic AEs - vaccination 2 | 6 | 3
  Serious AEs : All AEs - vaccination 1 | 0 | 1
  Serious AEs : All AEs - vaccination 2 | 1 | 1
  Serious AEs : Local AEs - vaccination 1 | 0 | 0
  Serious AEs : Systemic AEs - vaccination 1 | 0 | 1
  Serious AEs : Local AEs - vaccination 2 | 0 | 0
  Serious AEs : Systemic AEs - vaccination 2 | 1 | 1

5. Secondary Outcome: Evaluation of Residual LT in the Patch and on the Skin at the Patch Site Post-wear
Time Frame: 1 month
Population: Summary statistics are only shown for the LT Group in a protocol pre-defined subset of subjects, results for the Placebo Group were below the Limit of detection in all cases
Measure: Mean (Standard Deviation); unit: nanograms (ng)
Arm/Group | Group 1: 37.5 µg LT Patch
Number analyzed (Participants) | 22
nanograms (ng)
  Residual LT in the Patch (ng LT) | 15893 (6980)
  Residual LT in the Swab (ng LT) | 7231 (2939)
  Estimate of LT Delivered (ng LT) | 14376 (7609)

6. Secondary Outcome: Evaluation of LT-specific Immune Responses One-year After Original Treatment Regimen in LT Patch Group
Description: GMT
Time Frame: 13 months
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | Group 1: 37.5 µg LT Patch
Number analyzed (Participants) | 76
GMT
  GMT LT IgG - Day 380 | 1653.7 [1377.9 to 1984.8]
  GMT LT IgA - Day 380 | 122.3 [98.3 to 152.1]

7. Secondary Outcome: Evaluation of LT-specific Immune Responses One Year After Original Treatment Regimen in LT Patch Group
Description: GMFR
Time Frame: 13 months
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: 37.5 µg LT Patch
Number analyzed (Participants) | 76
ratio
  GMFR LT IgG - Day 380 | 3.8 [3.0 to 4.9]
  GMFR LT IgA - Day 380 | 2.4 [1.8 to 3.3]

8. Secondary Outcome: Evaluation of LT-specific Immune Responses One Year After Original Treatment Regimen in LT Patch Group
Description: SCR
Time Frame: 13 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: 37.5 µg LT Patch
Number analyzed (Participants) | 76
percentage of participants
  SCR LT IgG - Day 380 | 67.1 [54.9 to 77.9]
  SCR LT IgA - Day 380 | 38.6 [27.2 to 51.0]

ADVERSE EVENTS:
Arm/Group | Group 1: 37.5 µg LT Patch | Group 2: 0 µg LT Patch (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/81 | 2/39
Other Adverse Events (participants affected / at risk) | 79/81 | 32/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 37.5 µg LT Patch (N=81) | Group 2: 0 µg LT Patch (Placebo) (N=39)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 37.5 µg LT Patch (N=81) | Group 2: 0 µg LT Patch (Placebo) (N=39)
Diarrhoea (Gastrointestinal disorders) | 11 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 4
Blood glucose increased (Investigations) | 6 | 3
Haemoglobin decreased (Investigations) | 3 | 2
Protein urine present (Investigations) | 4 | 3
Application site discolouration (Injury, poisoning and procedural complications) | 62 | 5
Application site erythema (Injury, poisoning and procedural complications) | 72 | 14
Application site oedema (Injury, poisoning and procedural complications) | 11 | 0
Application site pain (Injury, poisoning and procedural complications) | 22 | 3
Application site pruritus (Injury, poisoning and procedural complications) | 72 | 8
Application site rash (Injury, poisoning and procedural complications) | 77 | 5
Malaise (General disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other